CLINICAL TRIAL: NCT06221410
Title: Investigating the Impact of Funny Scenario-Based Learning and Mind Mapping Methods on Undergraduate Students' Motivation to Learn Medical Terminology
Brief Title: Motivation in Learning Medical Terminology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, PARISA HADAVİBAVİLİ, Lecturer, Sakarya University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SAU-FHS-PHB-1
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Education; Medical Terminology Education
Keywords: Nursing Terminology; Education; Nursing Education; Active Learning

STUDY DESIGN:
Intervention Model Description: The participants were divided into three groups based on their preferences. Through this mechanism, they were able to cultivate a sense of responsibility and a sense of ownership in their educational journey.
  Specifically, students who engage in funny scenario-based education prefer to collaborate with peers who share similar interests and learning styles, which makes preparing scenarios more enjoyable.
  Meanwhile, in the mind-mapping groups, students draw on their creative skills to deconstruct and assimilate unfamiliar terms, utilizing their sense of humor and artistic competencies.
  The control group will only receive traditional teaching methods (PowerPoint). After the study, the control group will also experience "Funny Scenario-Based Learning" and "Mind Mapping."
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study was administered by two investigators. A traditional classroom teaching method was employed by the first investigator as a lecturer. the lecturer investigator administered both pre- and post-test scales to students. The second investigator was blinded to the group assignments of the students, ensuring unbiased data collection. The investigator was responsible for preparing and entering the data into SPSS for subsequent analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): The control group will only receive traditional teaching methods (PowerPoint).
- Funny Scenario-Based Group (Experimental): The "Funny Scenario-Based" approach is an educational approach where humor is integrated with scenario-based learning. Using this teaching strategy, comedic elements are incorporated into realistic or hypothetical scenarios to engage students and make learning more fun.
  In such scenarios, students may encounter a wide range of characters, situations, and challenges designed to entertain and engage students with different types of medical terms. It is common to incorporate humor into the educational process, helping to maintain educational relevance while appealing to the student's sense of enjoyment.
  Interventions: Other: Alternative teaching method: Funny Scenario-Based Education
- Mind-mapping Group (Experimental): The term "Mind-mapping Group" refers to a collaborative educational setting in which students use mind-mapping as an instructional strategy. A mind map is a visual thinking tool that involves diagramming tasks, words, concepts, or items that are related to and arranged around a central concept.
  Interventions: Other: Alternative teaching method: Mind-mapping Education

INTERVENTIONS:
Other: Alternative teaching method: Funny Scenario-Based Education — A humorous scenario is written and performed by students as part of this alternative educational intervention. The engaging approach facilitates both a deeper understanding of complex medical terminology and adds a sense of humor and fun to the learning process.
  Approximately 5 to 10 students will participate in each small group. A group size will be determined based on the voluntary interest and willingness of the students. These dynamic teams will provide students with opportunities to collaborate, enhance peer interaction, and cultivate soft skills such as communication and teamwork, all while having fun together.
  Arms: Funny Scenario-Based Group
Other: Alternative teaching method: Mind-mapping Education — As part of an alternative educational intervention, Mind-mapping Education encourages students to visually map out information, creating a graphic representation of their ideas and knowledge. Using such mind maps, students can see the connections and hierarchies in the information they are learning because they have a central idea with branches that denote related concepts, facts, and details.
  Arms: Mind-mapping Group

SUMMARY:
The aim of this study is to examine the impact of "Funny Scenario-Based Learning and Mind Mapping Methods" on undergraduate students' motivation to learn medical terminology. This research aims to assess the effectiveness of the specified methods in enhancing the English learning motivation of undergraduate students.

DETAILED DESCRIPTION:
Medical Terminology is a specialized language system that expresses the meanings and structures of terms used in the field of medicine. These terms are often of Latin and Greek origin and are widely used in medical documentation, communication, and education (Ismayilli Karakoc, 2020). The education of medical terminology is crucial for healthcare professionals to communicate effectively, understand medical documents, and have accurate knowledge about diseases. Additionally, the use of correct terms helps prevent errors (Antoniou et al., 2011).

Traditionally, textbooks and courses have played a fundamental role in teaching medical terminology to students, presenting structured content for learning basic terms (Sharipov et al., 2023). Nowadays, active methods used in medical terminology education include Flashcards, Online Resources and Applications, Scenario-Based Learning, and Mind Mapping (Alizadeh et al., 2021; Grezes & Decety, 2001; Hsu & Chen, 2023; Liu et al., 2017).

According to the literature, students' motivation has a significant impact on language education. Motivated students show more participation in classes, dedicate more time to the learning process, and achieve higher success (Grezes & Decety, 2001). Medical terminology education is especially important for nursing and midwifery students. Studies suggest that using correct terms in these professions ensures effective communication with patients and the accurate execution of treatment processes (Stedman, 2005).

In this study, students studying medical terminology at the Faculty of Health Sciences were evaluated for their learning motivation. The study population consists of students in the 2nd year of the Nursing and Midwifery Department at Sakarya University Faculty of Health Sciences between October 2023 and January 2024. This study is based on the voluntary participation of students.

The participants were divided into three groups based on their preferences. In addition to the traditional teaching methods (PowerPoint), one group will receive medical terminology English training through the "Funny Scenario-Based Learning" method, while the other group will receive training through the "Mind Mapping" method. Through this mechanism, they were able to cultivate a sense of responsibility and a sense of ownership in their educational journey. Consequently, it is anticipated that such autonomy could boost their motivation and engagement, potentially enhancing their educational performance.

Specifically, students who engage in funny scenario-based education prefer to collaborate with peers who share similar interests and learning styles, which makes preparing scenarios more enjoyable. A self-directed grouping likely fosters an environment of idea exchange, mutual encouragement, and collaborative assistance, resulting in a synergistic and supportive learning culture. As a result of peer support, students may be motivated by peer recognition, receive constructive feedback, and experience social interaction.

Meanwhile, in the mind-mapping groups, students draw on their creative skills to deconstruct and assimilate unfamiliar terms, utilizing their sense of humor and artistic competencies. As a result of this approach, students are required to engage actively with the content, allowing them to encode information in a creative and effective way.

The control group will only receive traditional teaching methods (PowerPoint). After the study, the control group will also experience "Funny Scenario-Based Learning" and "Mind Mapping."

The researchers will use the Scale of English Learning Motivation for Students Studying in the Faculty of Health Sciences as a pre-test and post-test for data collection.

The motivation levels of all three groups will be evaluated both before and after using the "English Learning Motivation Scale." Data collection tools include:

1. Student Information Questionnaire: This questionnaire consists of approximately 10 questions, capturing students' identifying information, including sociodemographic and academic details.
2. Scale of English Learning Motivation for Students in the Faculty of Health Sciences: This scale, developed by DEMİR and HAMARAT in 2022, comprises 14 items divided into three sub-dimensions (intrinsic motivation with 5 items, extrinsic (instrumental) motivation with 5 items, and integrative motivation with 4 items). All items on the scale are arranged in a five-point Likert scale ranging from "completely disagree" to "completely agree." The scoring of items on the scale is done on a Likert scale of 1 = definitely disagree to 5 = definitely agree. The evaluation of scores is based on the sum of item scores obtained from each factor. The scores obtained from each dimension of the scale can be ranked as follows: "Intrinsic motivation" and "Extrinsic motivation" factors can range from 5 to 25, while the "Integrative motivation" factor can range from 4 to 20. The total of the scale cannot be found by adding up the total scores because the scale is not a summation. A higher score obtained from any dimension indicates effectiveness in learning motivation. Additionally, there are no items reversed in the scale, and all items are formulated with positive expressions.

ELIGIBILITY:
Inclusion Criteria:

* Being a second-year student at Sakarya University's Faculty of Health Sciences.
* The first time taking a medical terminology course.
* An English second language speaker.

Exclusion Criteria:

* Refusing to participate in the research.
* Being a native English speaker.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-29 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
The aim of this study is determined as "Investigating the Impact of Funny Scenario-Based Learning and Mind Mapping Methods on Undergraduate Students' Motivation to Learn Medical Terminology." | 14 weeks
  In this study, students studying medical terminology at the Faculty of Health Sciences were evaluated for their learning motivation. The study population consists of students in the 2nd year of the Nursing and Midwifery Department at Sakarya University Faculty of Health Sciences between October 2023 and January 2024. The participants were divided into three groups based on their preferences. The researchers will use the Scale of English Learning Motivation for participants. The motivation levels of all three groups will be evaluated both before and after using the "English Learning Motivation Scale."

CONTACTS AND LOCATIONS:
Locations (1):
- Parisa Hadavi Bavili, Sakarya, Turkey (Türkiye)